CLINICAL TRIAL: NCT04166760
Title: Metabolic Effects of Whey Compounds in Patients With Diabetes Mellitus Type 2.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAKE4
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHE (regular whey protein) (Active Comparator): Regular whey protein. The intervention will be ingested 30 min. prior to an OGTT (3 hours). The intervention will also be ingested 30 min prior to breakfast and dinner for 2 days in the patient's own environment.
  Interventions: Dietary Supplement: WHE
- speWHE (specific whey protein compound) (Experimental): Specific whey protein compound. The intervention will be ingested 30 min. prior to an OGTT (3 hours). The intervention will also be ingested 30 min prior to breakfast and dinner for 2 days in the patient's own environment.
  Interventions: Dietary Supplement: speWHE

INTERVENTIONS:
Dietary Supplement: speWHE — 25 gram of a specific whey fraction (confidential)
  Arms: speWHE (specific whey protein compound)
Dietary Supplement: WHE — 25 gram protein of a regular whey compound
  Arms: WHE (regular whey protein)

SUMMARY:
The main objective of our study is to investigate the metabolic effects of a i) ordinary whey protein (WHE) and ii) a specific whey protein fraction (speWHE) when the interventions are ingested by patients with type 2 diabetes 30 minutes prior to an oral glucose tolerance test (OGTT). We will also investigate the glucose response when the patients ingest the interventions at home in their own environment 30 minutes before breakfast and dinner (2days) and also monitor glucose levels without interventions (2 days).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type 2 diabetes (T2D) diagnosis
* No medical treatment or metformin/sulfonylureas(SU) alone in the treatment of T2D
* No daily use of protein drinks
* Hba1c between 40 mmol/mol and 69 mmol/mol
* 20 kg/m2 < BMI < 35 kg/m2
* Screening blood test: 1200 pmol/l > C-peptid > 370 pmol/l

Exclusion Criteria:

* Other diabetes medication than metformin/SU (e.g. insulin, GLP-1 analog, DPP-4 inhibitor, SGLT2-inhibitor)
* Affected screening blood test assessed by the primary investigator(PI)/sponsor
* Does not understand or speak danish
* Milk allergy
* PI finds the patient not fit (e.g. mental illness, too nervous or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Difference in iAUC for insulin between WHE and speWHE | OGTT, 3 hours.
  Difference in iAUC for insulin between WHE and speWHE

SECONDARY OUTCOMES:
Differences in iAUC and concentration differences for GIP | OGTT 3 hours
Differences in iAUC and concentration differences for GLP-1 | OGTT 3 hours
Differences in iAUC and concentration differences for glucagon | OGTT 3 hours
Differences in iAUC and concentration differences for glucose | OGTT 3 hours
Differences in iAUC and concentration differences for C-peptid | OGTT 3 hours
Differences in iAUC and concentration differences for FFA | OGTT 3 hours
Activity measurements | 5 days
continuous glucose measurement (CGM) | 5 days
  CGM with time in normal range 4-10 mmol/l, peak after a meal, AUC in the days with the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jessen, Professor, Study Director — Medicinsk forskningslaboratorium for Diabetes og Hormonsygdomme og Steno Diabetes Center Aarhus (M-lab), Aarhus universitetshospital
Locations (1):
- Medicinsk forskningslaboratorium for Diabetes og Hormonsygdomme og Steno Diabetes Center Aarhus (M-lab), Aarhus universitetshospital, Aarhus, Denmark